CLINICAL TRIAL: NCT00708370
Title: An Outcome Research on the Impact of a Disease Management Program (COACH) on the Attainment of Better Cardiovascular Risk Control in Dyslipidemic Patients at Primary Care Centers (DISSEMINATE).
Brief Title: A Study to Evaluate the Efficacy of a Counselling and Advisory Care for Health (COACH) Program in Dyslipidemic Patients.
Acronym: DISSEMINATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A2581162
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Dyslipidemia
Keywords: Interventional; Non-drug; Disease Management Program; Cardiovascular Risk Control; Dyslipidemias; Primary Care Centers
MeSH Terms: conditions — Dyslipidemias | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- COACH (Active Comparator)
  Interventions: Other: COACH
- Standard Care (Placebo Comparator)
  Interventions: Other: No intervention for placebo

INTERVENTIONS:
Other: COACH — COACH Nurse will provide health tele-counselling to patients randomized to COACH arm fortnightly for 24 weeks.
  Other Names: COACH plus Standard Care
  Arms: COACH
Other: No intervention for placebo — There will be no COACH health tele-counselling to patients randomized to Standard Care arm.
  Other Names: Placebo
  Arms: Standard Care

SUMMARY:
This study is a local PCO sponsored, interventional, non-drug study to evaluate the efficacy of a health tele-counselling program in reducing cardiovascular risk in dyslipidemic patients.

DETAILED DESCRIPTION:
Educational / Counseling

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are newly diagnosed with dyslipidemias.
2. Subjects must be lipid drug naive and eligible for statin therapy.

Exclusion Criteria:

1. Subjects who cannot be contacted by telephone or handphone.
2. Subjects with uncontrolled primary hypothyroidism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Percentage (%) change from baseline to week 24 in serum LDL-C levels. | 24 weeks from Baseline

SECONDARY OUTCOMES:
Subjects' lifestyle modification as assessed by the incidence and frequency of smoking, consumption of foods high in salt, sugar and/or fat content, alcohol consumption, and exercise habits at baseline and weeks 24 and 36. | 24 and 36 weeks from Baseline
Percentage (%) change from baseline in serum LDL-C (week 36), TC (week 24 and 36), HDL-C (week 24 and 36), TG (week 24 and 36) and TC/HDL-C ratio (week 24 and 36). | 24 and 36 weeks from Baseline
Subjects' satisfaction with the Health Booklet and the COACH program after 24 weeks. | 24 weeks from Baseline
Absolute change in SBP and DBP from baseline to weeks 24 and 36. | 24 and 36 weeks from Baseline
Percentage (%) change in Framingham CHD risk score from baseline to weeks 24 and 36. | 24 and 36 weeks from Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- Malaysia (20):
  - Pfizer Investigational Site, Jitra, Kubang Pasu, Kedah
  - Pfizer Investigational Site, Kulim, Kedah
  - Pfizer Investigational Site, Sik, Kedah
  - Pfizer Investigational Site, Kubang Kerian, Kelantan
  - Pfizer Investigational Site, Cheras, Kuala Lumpur
  - Pfizer Investigational Site, Kuala Lumpur, Kuala Lumpur
  - Pfizer Investigational Site, Kampung Baharu Nilai, Negeri Sembilan
  - Pfizer Investigational Site, Tampin, Negeri Sembilan
  - Pfizer Investigational Site, Bagan Serai, Perak
  - Pfizer Investigational Site, Lenggong, Perak
  - Pfizer Investigational Site, Slim River, Perak
  - Pfizer Investigational Site, Kapar, Selangor
  - Pfizer Investigational Site, Petaling Jaya, Selangor
  - Pfizer Investigational Site, Puchong, Selangor
  - Pfizer Investigational Site, Sungai Buloh, Selangor
  - Pfizer Investigational Site, Kampong Kemaman, Terengganu
  - Pfizer Investigational Site, Kerteh, Kemaman, Terengganu
  - Pfizer Investigational Site, Kuala Lumpur
  - Pfizer Investigational Site, Malacca
  - Pfizer Investigational Site, Shah Alam

REFERENCES:
- [Derived] Selvaraj FJ, Mohamed M, Omar K, Nanthan S, Kusiar Z, Subramaniam SY, Ali N, Karanakaran K, Ahmad F, Low WH; DISSEMINATE study group. The impact of a disease management program (COACH) on the attainment of better cardiovascular risk control in dyslipidaemic patients at primary care centres (The DISSEMINATE Study): a randomised controlled trial. BMC Fam Pract. 2012 Oct 10;13:97. doi: 10.1186/1471-2296-13-97. PMID 23046818